CLINICAL TRIAL: NCT03285997
Title: A Study to Evaluate the Efficacy and Safety of GC3110A in Healthy Infants From 6 Months to 35 Months of Age
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GC3110A_IF_P3
Record Dates: First submitted 2017-09-13; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Influenza Vaccine
Keywords: Quadrivalent Influenza Vaccines
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GC3110A (Experimental): One injection: Day 0 Two injection: Day 0 and Day 28
  Interventions: Biological: GC3110A
- GCFLU Pre-filled syringe inj. (Active Comparator): One injection: Day 0 Two injection: Day 0 and Day 28
  Interventions: Biological: GCFLU Pre-filled syringe inj.

INTERVENTIONS:
Biological: GC3110A — A single 0.5mL dose intramuscular injection
  Arms: GC3110A
Biological: GCFLU Pre-filled syringe inj. — A single 0.25mL dose intramuscular injection
  Arms: GCFLU Pre-filled syringe inj.

SUMMARY:
If study subject's legal guardians who decide voluntarily to participate the clinical trial, and sign the Informed Consent Formed, study subjects eligible for participating this trial protocol were assigned to test group or control group with the ratio of 4:1 and receiving the test or control drug 1 time or 2 times.

DETAILED DESCRIPTION:
1. Part 1 If study subject's legal guardians who decide voluntarily to participate the clinical trial, and sign the Informed Consent Form, study subjects eligible for participating this trial protocol were assigned to test group and receiving the test drug 1 time or 2 times.
2. Part 2 If study subject's legal guardians who decide voluntarily to participate the clinical trial, and sign the Informed Consent Formed, study subjects eligible for participating this trial protocol were assigned to test group or control group with the ratio of 4:1 and receiving the test or control drug 1 time or 2 times.

The investigator will evaluate the efficacy and safety of the test product while clinical trial.

Blood samples will be collected at visit 1 and visit 5 for immunogenicity evaluation. The study subject and their legal guardians will be educated to daily record AEs after vaccination on the patient diary to evaluate the safety.

At visit1, blood samples will be collected from randomized study subjects and investigational drug will be intramuscularly injected. However, those who had not been vaccinated with influenza vaccine, will re-visit and have the 2nd vaccination, 4~5 weeks after the 1st vaccination.

After 4~5 weeks since last vaccination, study subjects will visit and blood sample will be collected. And the serious adverse events occurred during 180 days after the final vaccination will be checked through the telephone visit.

The study subjects with 1 dose of vaccine will have 4 visits including Visit 1~2 and Visit 5~6. The study subjects with 2 dose of vaccine will have 6 visits including Visit 3~4.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants aged 6 month to 3 years.
2. Study subject was born at full term pregnancy(37 week)
3. Study subject who understand the details of this clinical trial, decide voluntarily to participate the trial, and signed the Informed Consent Form

Exclusion Criteria:

1. Those with a history of allergic reaction to eggs or chicken, the vaccine components
2. Those who had been ad ministered the influenza vaccine 6 months prior to the study drug vaccination
3. Those with immunologic impairment including immune deficiency disorders or family history about it.
4. Those with a history of Guillain-Barre syndrome
5. Those with a history of Down's syndrome or cytogenetic disorders
6. Those who would be ineligible to participate the study as follows: serious chronic disease
7. Hemophilia patients at risk of serious bleeding with intramuscular injection or those receiving anticoagulant therapy
8. Those who have active infection or who have fever higher than 38.0℃ within 72 hours prior to the dosing of study drug
9. Those who had been vaccinated with another vaccine within 28 days prior to the dosing of study drug or had a scheduled vaccination during the clinical trial period
10. Those who had received an immunosuppressant, immunity-modifying drug within 3 months prior to the dosing of study drug
11. Those who had received immunoglobulin or a blood-derived product within 3 months prior to the dosing of study drug or is scheduled to receive those products during the study period
12. Those who had taken antipyretic/analgesic/nonsteroidal antiinflammatory drugs within 4 hours prior to the dosing of study drug
13. Study subject who had participated in other clinical trial within 28 days prior to the study vaccination

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 260 (Estimated)
Dates: Start 2017-09-30 (Estimated); Primary Completion 2018-05-31 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate for HI antibody after final injection | Post-vaccination (Day 28 or 56)
  the percentage of study subjects with a pre-vaccination (Day 0) HI titer<1:10 and post-vaccination (Day 28) HI antibody titer≥1:40(Case1), or the percentage of study subjects with a pre-vaccination HI antibody titer≥1:10 and a minimum four-fold rise in post-vaccination HI antibody titer(Case 2)
Seroprotection rate for HI antibody after final injection | Post-vaccination (Day 28 or 56)

SECONDARY OUTCOMES:
GMT | Post-vaccination (Day 28 or 56)
  GMT(Geometric Mean Titer) of HI antibody titer before vaccination(Day 0) and after vaccination (Day 28)
GMR | Post-vaccination (Day 28 or 56)
  GMR(Geometric Mean Ratio) of HI antibody titer before vaccination(Day 0) and after vaccination (Day 28)

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic Univ.of Korea Seoul St.Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi UY, Kim KH, Lee KY, Kim JH, Kim CS, Eun BW, Kim HM, Kim DH, Song SE, Jo DS, Lee J, Ma SH, Kim KN, Kang JH. Active-controlled phase III study of an egg-cultivated quadrivalent inactivated split-virion influenza vaccine (GC3110A) in healthy Korean children aged 6-35 months. Vaccine. 2021 Apr 8;39(15):2103-2109. doi: 10.1016/j.vaccine.2021.03.005. Epub 2021 Mar 16. PMID 33736920